CLINICAL TRIAL: NCT03500224
Title: A Phase 1, Open-label, Single Intravenous Infusion Dose Study to Evaluate the Mass Balance, Pharmacokinetics, Metabolism, and Excretion of TAK-954 Containing Microtracer ([14C]-TAK-954) in Healthy Adult Male Subjects
Brief Title: A Study to Evaluate the Mass Balance, Pharmacokinetics (PK), Metabolism and Excretion of TAK-954 Containing Microtracer ([14C]-TAK-954) in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-954-1005; U1111-1202-5762 (Other: WHO); NL65503.056.18 (Registry Identifier: NL); 2018-001181-42 (EudraCT Number)
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-TAK-954 0.5 mg (Experimental): [14C]-TAK-954 0.5 milligram (mg), (containing approximately 1.5 microcurie [µCi] of radioactive tracer), administered as 60-minute infusion, intravenously, once on Day 1.
  Interventions: Drug: [14C]-TAK-954

INTERVENTIONS:
Drug: [14C]-TAK-954 — [14C]-TAK-954 intravenous infusion.

SUMMARY:
The purpose of this study is to determine the mass balance, routes of elimination and characterize the metabolic profiles of a single intravenous dose of [14C]-TAK-954, identify major circulating and excreted metabolites. This study will also determine the single-dose PK of total radioactivity, TAK-954 and its metabolites where possible.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-954. This study will assess the mass balance, metabolic profiles and routes of elimination of single intravenous dose of [14C]-TAK-954, and will determine the major circulating and excreted metabolites and single-dose PK of total radioactivity, TAK-954, THRX513466, and THRX 913682 in healthy male participants.

The study will enroll approximately 6 participants. All participants will receive a single dose of [14C]-TAK-954 0.5 mg on Day 1.

This single-center trial will be conducted in Netherlands. The overall time to participate in this study is approximately 6 to 7 weeks. Participants will make a final visit to the clinic 15 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Be a man aged 18 to 55 years, inclusive, at the screening visit.
2. Have a body mass index (BMI) greater than or equal to (>=) 18 and less than or equal to (<=) 30 kilogram per square meter (kg/m^2) and a body weight greater than (>) 50 kilogram (kg) at the screening visit.
3. Be a nonsmoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months before administration of the initial dose of trial drug.
4. Meet the following birth control requirements:

   * Is a male participant who is sterile or agrees to use an appropriate method of contraception, including a condom, from the first dose of study drug until 30 days after the last dose of study drug. No restrictions are required for a vasectomized male participant provided that the participant is at least 1 year postbilateral vasectomy procedure before the first dose of study drug. A male participant whose vasectomy procedure was performed less than 1 year before the first dose of study drug must follow the same restrictions as a nonvasectomized man. Appropriate documentation of surgical procedures should be provided.
   * Is a male participant who agrees to not donate sperm from trial drug administration on the first day of the first dose until 30 days after the last dose of study drug.

Exclusion Criteria:

1. Has total 14C radioactivity measured by accelerator mass spectrometry in plasma (during screening) exceeding 14C/12C ratio 1.1E-12.
2. Participated in any study with a radiation dose above 0.1 millibecquerel (MBq) or radiation burden above 0.1 millisievert (mSv) within 1 year before screening.
3. Was exposed to significant radiation (example, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months before check-in.
4. Irregular defecation pattern (less than once per 2 days).
5. Has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to beer 354 milliliter [mL]/12 ounce [oz], wine 118 mL/4 oz, or distilled spirits 29.5 mL/1 oz).
6. Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
7. Has a substance abuse disorder.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- PRAHS, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the Netherlands from 30 April 2018 to 01 June 2018.
Pre-assignment Details: Healthy participants were enrolled to receive a single 60-minute intravenous infusion of 0.5 milligram (mg) TAK-954 containing a microtracer of [14C]-TAK-954.
Groups:
- [14C]-TAK-954 0.5 mg: [14C]-TAK-954 0.5 mg (containing approximately 1.5 µCi) of radioactive tracer administered as a 60-minute infusion, intravenously, once on Day 1.
Period: Overall Study
Arm/Group | [14C]-TAK-954 0.5 mg
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 6
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 76.37 (8.694)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 177.2 (7.78)
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.2 (1.72)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Percentage of Administered Radioactivity Recovered in Urine
Time Frame: Day 1 pre-dose and at multiple time points (up to 264, 312, and 336 hours) post-dose
Population: The pharmacokinetic (PK) analysis set included all the participants of safety analysis set with sufficient concentration data to facilitate the derivation of at least 1 PK parameter from the concentration time data. The PK analysis set where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: percentage of radioactive dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of radioactive dose
  0 to 264 hours | 55.4 (3.2)
  0 to 312 hours: number analyzed (Participants) | 3
  0 to 312 hours | 56.8 (3.2)
  0 to 336 hours: number analyzed (Participants) | 2
  0 to 336 hours | 55.1 (0.4)

2. Primary Outcome: Cumulative Percentage of Administered Radioactivity Recovered in Feces
Time Frame: Day 1 pre-dose and at multiple time points (up to 264, 312, and 336 hours) post-dose
Population: The PK analysis set included all the participants of safety analysis set with sufficient concentration data to facilitate the derivation of at least 1 PK parameter from the concentration time data. The PK analysis set where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: percentage of radioactive dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of radioactive dose
  0 to 264 hours | 28.8 (2.5)
  0 to 312 hours: number analyzed (Participants) | 3
  0 to 312 hours | 30.3 (2.5)
  0 to 336 hours: number analyzed (Participants) | 2
  0 to 336 hours | 30.0 (3.5)

3. Primary Outcome: Cumulative Percentage of Radioactivity in Urine and Feces Combined
Time Frame: Day 1 pre-dose and at multiple time points (up to 264, 312, and 336 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of radioactive dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of radioactive dose
  0 to 264 hours | 84.1 (5.3)
  0 to 312 hours: number analyzed (Participants) | 3
  0 to 312 hours | 87.0 (4.6)
  0 to 336 hours: number analyzed (Participants) | 2
  0 to 336 hours | 85.1 (3.9)

4. Primary Outcome: Normalized Recovery as Percentage of Dose for TAK-954 and TAK-954 Metabolites in Urine and Feces Combined
Description: Percentage of dose recovered for TAK-954 and its metabolites derived from 0-168 hour sampling was normalized for 100% recovery.
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: PK analysis set: All participants of safety set with sufficient data to facilitate at least 1 PK parameter from concentration time data. Single value is available for Metabolite (M) 16, M4, and M5 because they co-eluted under chromatographic conditions. Single sampling method used across participants, therefore there was no measure of dispersion.
Measure: Number; unit: percentage of dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of dose
  M1 | 3.0
  M3 | 13.6
  M14 | 4.3
  M4, M5, and M16 | 5.0
  M17 | 1.6
  M7 | 0.5
  M9 | 0.6
  M10 | 1.0
  TAK-954 | 58.0

5. Primary Outcome: Normalized Recovery as Percentage of Dose for TAK-954 and TAK-954 Metabolites in Urine
Description: as for outcome 4
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 4
Measure: Number; unit: Percentage of dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
Percentage of dose
  M1 | 3.0
  M3 | 4.8
  M14 | 4.3
  M5, M4, and M16 | 1.6
  M17 | 0.8
  M9 | 0.6
  M10 | 0.5
  TAK-954 | 44.3

6. Primary Outcome: Normalized Recovery as Percentage of Dose for TAK-954 and TAK-954 Metabolites in Feces
Description: as for outcome 4
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 4
Measure: Number; unit: percentage of dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of dose
  M3 | 8.8
  M5, M4, and M16 | 3.4
  M17 | 0.8
  M7 | 0.5
  M10 | 0.5
  TAK-954 | 13.7

7. Primary Outcome: Mean Percent of Total Radioactivity in Plasma for TAK-954 and TAK-954 Metabolites
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The PK analysis set included all the participants of safety analysis set with sufficient concentration data to facilitate the derivation of at least 1 PK parameter from the concentration time data. Data is reported for TAK-954. Data for metabolites are not reported because none exceeded greater than (>) 6% of the total plasma radioactivity.
Measure: Mean (Standard Deviation); unit: percentage of total radioactivity
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of total radioactivity | 74.28 (8.18)

8. Primary Outcome: Cumulative Percentage of Dose Excreted in Urine for TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 264, 312, and 336 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of dose
  0 to 264 hours | 31.33 (3.29)
  0 to 312 hours: number analyzed (Participants) | 3
  0 to 312 hours | 29.73 (4.14)
  0 to 336 hours: number analyzed (Participants) | 2
  0 to 336 hours | 27.35 (0.35)

9. Primary Outcome: Cumulative Percentage of Dose Excreted in Feces for TAK-954
Description: The cumulative percentage of dose excreted in feces as TAK-954 derived from 0-168 hour sampling was normalized for 100% recovery.
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The PK analysis set included all the participants of safety analysis set with sufficient concentration data to facilitate the derivation of at least 1 PK parameter from the concentration time data. Single sampling method used across participants, therefore there was no measure of dispersion.
Measure: Number; unit: percentage of dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of dose | 13.7

10. Primary Outcome: Mean Concentration of Total Radioactivity in Whole Blood and Plasma [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram equivalent/milliliter(ng eq/mL)
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
nanogram equivalent/milliliter(ng eq/mL)
  Whole Blood: 0.00 minute | NA (NA) — Data were not reported because none of the values were above lower limit of quantification (LLOQ).
  Whole Blood: 0.50 minute | 5.15 (0.908)
  Whole Blood: 1 hour | 5.87 (1.26)
  Whole Blood: 1.5 hour | 2.88 (0.523)
  Whole Blood: 2 hour | 2.40 (0.418)
  Whole Blood: 3 hour | 2.05 (0.349)
  Whole Blood: 4 hour | 2.09 (0.407)
  Whole Blood: 6 hour | 1.79 (0.385)
  Whole Blood: 12 hour | 1.40 (0.217)
  Whole Blood: 24 hour | 0.923 (0.114)
  Whole Blood: 36 hour | 0.583 (0.0874)
  Whole Blood: 72 hour | 0.232 (0.0530)
  Whole Blood: 96 hour | 0.140 (0.0420)
  Whole Blood: 120 hour | 0.0953 (0.0292)
  Whole Blood: 144 hour | 0.0695 (0.0211)
  Whole Blood: 168 hour | 0.0449 (0.0363)
  Whole Blood: 192 hour: number analyzed (Participants) | 5
  Whole Blood: 192 hour | 0.0352 (0.0332)
  Whole Blood: 216 hour | 0.0268 (0.0301)
  Whole Blood: 240 hour | 0.0246 (0.0273)
  Whole Blood: 264 hour | 0.00940 (0.0230)
  Whole Blood: 288 hour: number analyzed (Participants) | 3
  Whole Blood: 288 hour | NA (NA) — Data were not reported because none of the values were above LLOQ.
  Whole Blood: 312 hour: number analyzed (Participants) | 2
  Whole Blood: 312 hour | NA (NA) — Data were not reported because none of the values were above LLOQ.
  Whole Blood: 336 hour: number analyzed (Participants) | 2
  Whole Blood: 336 hour | NA (NA) — Data were not reported because none of the values were above LLOQ.
  Plasma: 0.00 minute | NA (NA) — Data were not reported because none of the values were above LLOQ.
  Plasma: 0.50 minute | 5.74 (1.72)
  Plasma: 1 hour | 6.29 (1.22)
  Plasma: 1.5 hour | 3.06 (0.528)
  Plasma: 2 hour | 2.59 (0.566)
  Plasma: 3 hour | 2.27 (0.495)
  Plasma: 4 hour | 2.17 (0.437)
  Plasma: 6 hour | 1.77 (0.433)
  Plasma: 12 hour | 1.34 (0.209)
  Plasma: 24 hour | 0.983 (0.104)
  Plasma: 36 hour | 0.601 (0.0567)
  Plasma: 48 hour | 0.443 (0.0478)
  Plasma: 72 hour | 0.271 (0.0502)
  Plasma: 96 hour | 0.169 (0.0368)
  Plasma: 120 hour | 0.123 (0.0378)
  Plasma: 144 hour | 0.0907 (0.0276)
  Plasma: 168 hour | 0.0689 (0.0264)
  Plasma: 192 hour | 0.0552 (0.0163)
  Plasma: 216 hour | 0.0480 (0.0131)
  Plasma: 240 hour | 0.0486 (0.0175)
  Plasma: 264 hour | 0.0407 (0.0114)
  Plasma: 288 hour: number analyzed (Participants) | 3
  Plasma: 288 hour | 0.0429 (0.0166)
  Plasma: 312 hour: number analyzed (Participants) | 2
  Plasma: 312 hour | 0.0413 (0.00559)
  Plasma: 336 hour: number analyzed (Participants) | 2
  Plasma: 336 hour | 0.0349 (0.00700)

11. Primary Outcome: Cmax: Maximum Observed Plasma and Whole Blood Concentrations of Radioactivity for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: The PK analysis set included all the participants of safety analysis set with sufficient concentration data to facilitate the derivation of at least 1 PK parameter from the concentration time data.
Measure: Geometric Mean (Full Range); unit: ng eq/mL
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
ng eq/mL
  Plasma | 6.28 [4.99 to 8.93]
  Whole Blood | 5.78 [4.10 to 7.75]

12. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-954 and TAK-954 Metabolites
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: The PK analysis set included all the participants of safety analysis set with sufficient concentration data to facilitate the derivation of at least 1 PK parameter from the concentration time data. PK data for TAK-954 metabolite THRX913682 could not be evaluated since its plasma levels were less than (<) lower limit of quantification.
Measure: Geometric Mean (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL)
  TAK-954 | 5.91 [5.08 to 7.79]
  THRX-513466 | 0.0143 [0.00998 to 0.0182]

13. Primary Outcome: AUClast: Area Under the Plasma and Whole Blood Radioactivity-time Curve From Time 0 to the Time of the Last Quantifiable Radioactivity for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Geometric Mean (Full Range); unit: h*ng eq/mL
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
h*ng eq/mL
  Plasma | 83.6 [74.4 to 89.5]
  Whole Blood | 75.4 [64.9 to 87.1]

14. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-954 and TAK-954 Metabolites
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: The PK analysis set included all the participants of safety analysis set with sufficient concentration data to facilitate the derivation of at least 1 PK parameter from the concentration time data. PK data for TAK-954 metabolite THRX913682 could not be evaluated since its plasma levels were < lower limit of quantification.
Measure: Geometric Mean (Full Range); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
hour*nanogram per milliliter (h*ng/mL)
  TAK-954 | 55.4 [46.2 to 66.5]
  THRX-513466 | 0.0371 [0.00739 to 0.156]

15. Primary Outcome: AUC∞: Area Under the Plasma and Whole Blood Radioactivity-time Curve From Time 0 to Infinity for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Geometric Mean (Full Range); unit: h*ng eq/mL
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
h*ng eq/mL
  Plasma | 87.2 [76.9 to 94.0]
  Whole Blood | 79.0 [67.6 to 92.1]

16. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-954 and TAK-954 Metabolites
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: The PK analysis set. PK data for metabolites could not be evaluated since metabolites were < lower limit of quantification and apparent terminal elimination portion of the concentration-time curve could not be characterized.
Measure: Geometric Mean (Full Range); unit: h*ng/mL
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
h*ng/mL | 55.7 [46.4 to 66.8]

17. Primary Outcome: Tmax: Time to Reach the Maximum Plasma and Whole Blood Radioactivity for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
hour
  Plasma | 1.00 [0.50 to 1.02]
  Whole Blood | 1.00 [0.55 to 1.02]

18. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-954 and TAK-954 Metabolites
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: The PK analysis set included all the participants of safety analysis set with sufficient concentration data to facilitate the derivation of at least 1 PK parameter from the concentration time data. PK data for TAK-954 metabolite (THRX913682) could not be evaluated since metabolites were < lower limit of quantification.
Measure: Geometric Mean (Full Range); unit: hour
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
hour
  TAK-954 | 1.00 [1.00 to 1.02]
  THRX-513466 | 1.00 [0.55 to 1.02]

19. Primary Outcome: t1/2z: Terminal Disposition Phase Half-life of Radioactivity in Plasma and Whole Blood for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Geometric Mean (Full Range); unit: hour
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
hour
  Plasma | 70.0 [57.9 to 89.9]
  Whole Blood | 46.4 [30.2 to 73.6]

20. Primary Outcome: t1/2z: Terminal Disposition Phase Half-life in Plasma for TAK-954 and TAK-954 Metabolites
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 16
Measure: Geometric Mean (Full Range); unit: hour
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
hour | 34.3 [23.1 to 47.0]

21. Primary Outcome: CL: Total Clearance After Intravenous Administration for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: No participant was analyzed since this outcome measure was not planned to be assessed but added in the protocol summary by error.
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 0

22. Primary Outcome: CL: Total Clearance of TAK-954 After Intravenous Administration of [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
L/h | 8.97 [7.49 to 10.8]

23. Primary Outcome: Vz: Volume of Distribution During the Terminal Disposition Phase After Intravenous Administration for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 21
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 0

24. Primary Outcome: Vz: Volume of Distribution During the Terminal Disposition Phase After Intravenous Administration for TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Geometric Mean (Full Range); unit: liter
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
liter | 444 [337 to 668]

25. Primary Outcome: Aet Urine: Amount of Total Radioactivity Excreted in Urine From Time 0 to Time t for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: microgram equivalent (mcg eq)
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
microgram equivalent (mcg eq) | 278 (16.2)

26. Primary Outcome: Aet Urine: Amount of Drug Excreted in Urine From Time 0 to Time t for TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
microgram (mcg) | 157 (16.4)

27. Primary Outcome: Aet Feces: Amount of Total Radioactivity Excreted in Feces From Time 0 to Time t for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg eq
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
mcg eq | 144 (12.9)

28. Primary Outcome: Fet Urine: Fraction of Drug Excreted in Urine From Time 0 to Time t for TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of dose | 31.3 (3.3)

29. Primary Outcome: Fet Urine: Fraction of Total Radioactivity Excreted in Urine From Time 0 to Time t for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of dose | 55.6 (3.2)

30. Primary Outcome: Fet Feces: Fraction of Radioactivity Excreted in Feces From Time 0 to Time t for [14C]-TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of dose | 28.8 (2.6)

31. Secondary Outcome: Ratio of Total Radioactivity in Whole Blood to Plasma
Time Frame: Day 1 pre-dose and at multiple time points (up to 264 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
ratio
  0.50 minute | 0.92 (0.13)
  1 hour | 0.93 (0.06)
  1.5 hour | 0.94 (0.09)
  2 hour | 0.94 (0.15)
  3 hour | 0.92 (0.17)
  4 hour | 0.96 (0.06)
  6 hour | 1.02 (0.14)
  12 hour | 1.04 (0.04)
  24 hour | 0.94 (0.07)
  36 hour | 0.97 (0.11)
  72 hour | 0.86 (0.08)
  96 hour | 0.82 (0.13)
  120 hour | 0.78 (0.12)
  144 hour | 0.79 (0.21)
  168 hour: number analyzed (Participants) | 4
  168 hour | 0.85 (0.16)
  192 hour: number analyzed (Participants) | 3
  192 hour | 1.17 (0.65)
  216 hour: number analyzed (Participants) | 3
  216 hour | 1.06 (0.37)
  240 hour: number analyzed (Participants) | 3
  240 hour | 1.04 (0.35)
  264 hour: number analyzed (Participants) | 1
  264 hour | 0.97 (NA) — Standard deviation could not be calculated since only one participant was analyzed.

32. Secondary Outcome: Ratio of AUC∞: Ratio of Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-954 to Total Radioactivity in Plasma TAK-954
Time Frame: Day 1 pre-dose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
ratio | 0.642 (0.0741)

33. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: Baseline up to Day 31
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of participants | 50.0

34. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) Leading to Discontinuation of [14C]-TAK-954
Time Frame: Baseline up to Day 15
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | [14C]-TAK-954 0.5 mg
Number analyzed (Participants) | 6
percentage of participants | 0.0

ADVERSE EVENTS:
Time Frame: A treatment-emergent adverse event (TEAE) are adverse events that started after the first dose of study drug and no more than 30 days (Day 31) after receiving the study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | [14C]-TAK-954 0.5 mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]-TAK-954 0.5 mg (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Head Discomfort (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT03500224/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT03500224/SAP_001.pdf